CLINICAL TRIAL: NCT03936257
Title: Evaluation of an Innovative BIO Formula Based on a New Whey Extraction Process on the Growth and Tolerance of Infants From 0 to 6 Months.
Brief Title: Effect of an Innovative BIO Formula Intake on Infant Growth and Tolerance From 0 to 6 Months
Acronym: TRUEGREEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Collaborators: Sodiaal International (Industry)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, Professor, Institut Pasteur de Lille
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2018-A00732-53
Record Dates: First submitted 2018-12-03; First posted 2019-05-03 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Child Development
MeSH Terms: interventions — Lactation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breast milk (Placebo Comparator): group receiving breastfeeding
  Interventions: Other: Breastfeeding
- infant formula conventional BIO (Active Comparator): infant formula with conventional whey BIO
  Interventions: Other: Conventional BIO Infant formula
- infant formula BIO TrueGreen (Active Comparator): infant formula with whey BIO TrueGreen
  Interventions: Other: TrueGreen BIO infant formula

INTERVENTIONS:
Other: Breastfeeding — Infants were breastfed during 3 months minimum. Data on growth and tolerance were collected. 10 out of 40 infants take a blood test to metabolome analysis
  Arms: Breast milk
Other: Conventional BIO Infant formula — Infant were fed during 6 months with a conventional BIO infant formula. Data on growth and tolerance were collected. 10 out of 40 infants take a blood test to metabolome analysis
  Arms: infant formula conventional BIO
Other: TrueGreen BIO infant formula — Infant were fed during 6 months with the TrueGreen BIO infant formula. Data on growth and tolerance were collected. 10 out of 40 infants take a blood test to metabolome analysis
  Arms: infant formula BIO TrueGreen

SUMMARY:
From birth to 5 months, milk is the essential and unique food of the newborn. The French National Nutrition Program (PNNS) recommends exclusive breastfeeding "up to 6 months and at least 4 months for a healthy benefit". However, only 36% of infants 0-6 months of age are exclusively breastfed worldwide. Some mothers choose to give infant formula to their baby in the first few months of life. This decision may be a personal choice or be imposed by pathophysiological situations.

The nutritional requirements of the infant are specific, which implies adequate nutrition. Infant formulas and follow-up formulas are therefore complex products, specially developed for a group of vulnerable consumers. In fact, the compositional and information requirements for infant formula are highly regulated.

This study, defined as a pilot study, proposes to evaluate the innovative "TrueGreen" BIO infant formula based on a new whey extraction method on the growth and tolerance of infants from 0 to 6 months compared to the conventional BIO infant formula. As no growth and tolerance data are currently available for this new TrueGreen BIO formula, this study aims to determine them.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 3 weeks
* Child followed by a general practitioner or pediatrician
* Informed consent form signed by the legal representatives of the subject
* Commitment of legal representatives to follow the constraints generated by the study
* Insured

Exclusion Criteria:

* Infant born prematurely before 37 weeks of amenorrhea
* Child allergic to cow's milk proteins
* Pathological pregnancy (hypertension, infection, gestational diabetes, etc.);
* Chronic or acute illness (metabolic or neuromuscular diseases, epilepsy, asthma, diabetes, digestive, renal, cardiac or haematological diseases);
* Incapacity for the legal representative(s) to understand or adhere to the protocol
* Subject involved in another clinical study or in an exclusion period from another study
* Legal representatives deprived of liberty
* Legal representatives in a position to judicial protection
* Weight of the subject according to age and sex, not included between the 3rd and the 97th percentile of the WHO Child Growth Standards
* Subject height according to age and sex, not between the 3rd and the 97th percentile of the WHO Child Growth Standards
* BMI of the subject according to age and sex, not included between the 3rd and the 97th percentile of the WHO Child Growth Standards
* Head circumference of the subject according to age and sex, not included between the 3rd and the 97th percentile of the WHO (World Health Organization) Child Growth Standards
* The investigator considers that the state of health or the concomitant treatments are not compatible with the good progress of the clinical study.

Ages: 1 Day to 21 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Evolution of growth of infants | from 0 to 6 months
  Weight in kilograms

SECONDARY OUTCOMES:
Height evolution of infants | from 0 to 6 months
  data in centimeters
BMI evolution of infants | from 0 to 6 months
  data in kg/m²
Head circumference evolution of infants | from 0 to 6 months
  data in centimeters
Number of colic per day | from 0 to 6 months
  Evaluation during 3 consecutives days every month.
Consistency of stool | from 0 to 6 months
  Evaluation during 3 consecutive days every month via Bristol scale.
  According to the bristol scale, seven types of stool are considered:
  Type 1: Separate hard lumps, like nuts (hard to pass) Type 2: Sausage-shaped, but lumpy Type 3: Like a sausage but with cracks on its surface Type 4: Like a sausage or snake, smooth and soft Type 5: Soft blobs with clear cut edges (easy to pass) Type 6: Fluffy pieces with ragged edges, a mushy stool Type 7: Watery, no solid pieces, entirely liquid
  The mean of stool type during 3 days is considered.
Number of regurgitation | from 0 to 6 months
  Evaluation during 3 consecutive days every month via Vandenplas scale.
  According to the Vandenplas scale, seven score are considered:
  0 0-2 episodes/day
  1. ≥3-≤5 of small volume
  2. >5 episodes of >1 coffee spoon
  3. >5 episodes of half of the feedings in < half of the feedings
  4. Continuous regurgitations of small volumes >30 min after each feeding
  5. Regurgitation of half to complete volume of a feeding in at least half of the feedings
  6. Regurgitation of the 'complete feeding' after each feeding
  The mean of score during 3 days is considered.
Number of wake up per night | from 0 to 6 months
  Evaluation during 3 consecutive days every month.
Total sleep time per day | from 0 to 6 months
  Time in hours. Evaluation during 3 consecutive days every month.
Plasma amino acid profile | between 3rd and 4th month
  Methods : Liquid Chromatography and Tandem Mass Spectrometry (LC / MS / MS) List of amino acids : Taurine, Aspartic acid, Threonine, Serine, Asparagine, Glutamine acid, Glutamine, Glycine, Alanine, Citrulline, Valine, Cystine, Methionine, Isoleucine, Leucine, Tyrosine, Phenylalanine, Beta aminoisobutyric acid, Ornithine, 1-Methyl-Histidine, Histidine, Lysine, 3-methyl-Histidine, Arginine, Hydroxyproline, Proline
Metabolomic analysis from plasma and urine samples | between 3rd and 4th month
  Non-targeted analysis : evaluation of all small molecules in biological system, such as amino acids, sugars, alcohols, sugar phosphates, amines, fatty acids, polar lipids, hormones and vitamins, as well as specialized metabolites, such as phenolic compounds, flavonoids, monoterpenes, sesquiterpenes, polyketides, alkaloids, including xenobiotics.
  Methods : Liquid Chromatography and Mass Spectrometry (LC / MS)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Lecerf, MD, Principal Investigator — Institut Pasteur de Lille - NutrInvest
Locations (1):
- NutrInvest - Institut Pasteur de Lille, Lille, Nord, France